CLINICAL TRIAL: NCT02422069
Title: Registry on Post Menopausal Osteoporosis in Gynecology Setting in Pakistan (REPOSE)
Brief Title: Study of Post Menopausal Osteoporosis (PMO) Among Gynecology Outpatients in Pakistan
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25212
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Study Population: Gynecology outpatients who meet eligibility criteria will be enrolled and evaluated for the presence of PMO at screening. Women diagnosed with PMO will complete an additional visit to document the prescribed management plan.

SUMMARY:
This observational study will provide an opportunity to document local patterns of susceptibility, patient profile, and usefulness of screening in postmenopausal patients coming to gynecology outpatient clinics in Pakistan. This will also capture the initial management of PMO in diagnosed patients. The information gathered will serve as a foundation for developing national guidelines on screening and management of PMO in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age 50 years or greater

Exclusion Criteria:

* Previously diagnosed osteoporosis, or receiving treatment for osteoporosis

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll gynecology outpatients in Pakistan who meet eligibility criteria for observation.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients diagnosed with PMO based upon dual-energy X-ray absorptiometry (DXA) results | Up to 12 months

SECONDARY OUTCOMES:
Use of various PMO treatment modalities | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Pakistan (4):
  - Islamabad
  - Karachi
  - Lahore
  - Rawalpindi